CLINICAL TRIAL: NCT01558427
Title: Salvage Treatment or Active Clinical Surveillance for Oligometastatic Prostate Cancer: a Randomized Phase II Trial
Brief Title: Non-systemic Treatment for Patients With Low-volume Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/156
Record Dates: First submitted 2012-03-12; First posted 2012-03-20 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active clinical surveillance (Experimental): Active monitoring of patients with low volume metastases with Prostate Specific Antigen (PSA) and sequential imaging.
  Interventions: Procedure: Surveillance
- Salvage treatment of metastases (Experimental): Surgical or radiotherapy treatment of metastases.
  Interventions: Procedure: Salvage treatment

INTERVENTIONS:
Procedure: Surveillance — Active clinical surveillance
  Arms: Active clinical surveillance
Procedure: Salvage treatment — Surgical removal of metastases, or stereotactic body radiotherapy of metastases.
  Arms: Salvage treatment of metastases

SUMMARY:
Prostate cancer patients diagnosed with a biochemical recurrence and limited metastases are conventionally treated with androgen deprivation therapy. However, in patients with limited metastatic load, the time to progression might be. Subsequently, active surveillance of these patients until progression might defer the start of androgen deprivation therapy (ADT) for several months to years. As an alternative, salvage treatment of the limited number of metastases with either surgery or radiotherapy might postpone the start of ADT even longer. The current trial hypothesizes that ADT might be deferred longer following salvage treatment as compared to active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of prostate cancer (PCa)
* Biochemical relapse of PCa following radical local prostate treatment
* N1 and M1a/b disease on imaging, with a combined maximum of 3 synchronous lesions.
* World Health Organization (WHO) performance state 0-1
* Exclusion of local relapse
* Age >=18 years old
* Signed informed consent

Exclusion Criteria:

* Serum testosterone level <50ng/ml
* Symptomatic metastases
* PSA rise while on active treatment with luteinizing hormone-releasing hormone (LHRH)-agonist, LHRH-antagonist, anti-androgen, maximal androgen blockade, oestrogen
* Previous treatment with cytotoxic agent for PCa
* Treatment during the past month with products known to influence Prostate Specific Antigen (PSA) levels (e.g. fluconazole, finasteride, corticosteroids,…)
* Disorder precluding understanding of trial information or informed consent

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Androgen deprivation therapy free survival. | From date of randomization until androgen deprivation therapy is started, assessed up to 2 years.
  Androgen deprivation therapy free survival will be calculated from randomization until androgen deprivation therapy is started.

SECONDARY OUTCOMES:
Quality of life questionnaire 1. | At 3, 6, 9, 12, 15, 18, 21, 24 months
  Questionnaire: European Organisation for Research and Treatment of Cancer Quality Of Life C30 (EORTC QLQ C30)
Quality of Life questionnaire 2. | At 3, 6, 9, 12, 15, 18, 21, 24 months
  Questionnaire: Short Form (36) Health Survey (SF36)
Quality of life questionnaire 3 | At 3, 6, 9, 12, 15, 18, 21, 24 months
  Questionnaire: EORTC QLQ PR25

CONTACTS AND LOCATIONS:
Overall Officials: Gert De Meerleer, PhD, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Deek MP, Van der Eecken K, Sutera P, Deek RA, Fonteyne V, Mendes AA, Decaestecker K, Kiess AP, Lumen N, Phillips R, De Bruycker A, Mishra M, Rana Z, Molitoris J, Lambert B, Delrue L, Wang H, Lowe K, Verbeke S, Van Dorpe J, Bultijnck R, Villeirs G, De Man K, Ameye F, Song DY, DeWeese T, Paller CJ, Feng FY, Wyatt A, Pienta KJ, Diehn M, Bentzen SM, Joniau S, Vanhaverbeke F, De Meerleer G, Antonarakis ES, Lotan TL, Berlin A, Siva S, Ost P, Tran PT. Long-Term Outcomes and Genetic Predictors of Response to Metastasis-Directed Therapy Versus Observation in Oligometastatic Prostate Cancer: Analysis of STOMP and ORIOLE Trials. J Clin Oncol. 2022 Oct 10;40(29):3377-3382. doi: 10.1200/JCO.22.00644. Epub 2022 Aug 24. PMID 36001857
- [Derived] Ost P, Reynders D, Decaestecker K, Fonteyne V, Lumen N, De Bruycker A, Lambert B, Delrue L, Bultijnck R, Claeys T, Goetghebeur E, Villeirs G, De Man K, Ameye F, Billiet I, Joniau S, Vanhaverbeke F, De Meerleer G. Surveillance or Metastasis-Directed Therapy for Oligometastatic Prostate Cancer Recurrence: A Prospective, Randomized, Multicenter Phase II Trial. J Clin Oncol. 2018 Feb 10;36(5):446-453. doi: 10.1200/JCO.2017.75.4853. Epub 2017 Dec 14. PMID 29240541
- [Derived] Ploussard G, Almeras C, Briganti A, Giannarini G, Hennequin C, Ost P, Renard-Penna R, Salin A, Lebret T, Villers A, Soulie M, de la Taille A, Flamand V. Management of Node Only Recurrence after Primary Local Treatment for Prostate Cancer: A Systematic Review of the Literature. J Urol. 2015 Oct;194(4):983-8. doi: 10.1016/j.juro.2015.04.103. Epub 2015 May 9. PMID 25963190
- [Derived] Decaestecker K, De Meerleer G, Ameye F, Fonteyne V, Lambert B, Joniau S, Delrue L, Billiet I, Duthoy W, Junius S, Huysse W, Lumen N, Ost P. Surveillance or metastasis-directed Therapy for OligoMetastatic Prostate cancer recurrence (STOMP): study protocol for a randomized phase II trial. BMC Cancer. 2014 Sep 15;14:671. doi: 10.1186/1471-2407-14-671. PMID 25223986
- See also: Related Info — http://www.uzgent.be